CLINICAL TRIAL: NCT04529954
Title: An Open-Label Extension Study to Investigate the Long-Term Safety, and Tolerability of Intracerebroventricular (ICV) Delivery of Valproate in Subjects With Focal Seizures, With Temporal Lobe Onset With or Without Secondary Generalization
Brief Title: Anti-Epilepsy Medication Valproate Administered Via ICV Route and Catheters and Pumps for CSF Infusion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Cerebral Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN100P.02
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label Safety (Experimental): Participants roll-over from DA071976 or CLN100P.02
  Interventions: Drug: Valproic Acid delivered to ICV

INTERVENTIONS:
Drug: Valproic Acid delivered to ICV — Valproic Acid delivered to ICV via an implantable pump and catheter system

SUMMARY:
This is a non-randomized open-label extension study for subjects having completed protocol DA071976 or CLN100P.01.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the DA07976 or CLN100P.01 Study
2. In the opinion of the investigator, if the subject were to be removed from study and associated therapy, subject would have worsening/increase in disabling seizures. Disabling refers to seizures that are severe enough to cause injuries, or significantly impair functional ability in domains including employment, psychosocial education and mobility.
3. Subject is taking currently approved AED medication(s) (but is not on valproate or divalproex sodium).
4. Subject has seizures that are distinct, stereotypical events that can be reliably counted, in the opinion of the Investigator, by the subject or caregiver.
5. Subject has hearing, vision, and physical abilities adequate to perform assessments, with or without corrective aids, including keeping a seizure and medication diary during study follow-up.
6. Subject understands study procedures and has voluntarily provided signed, informed consent in accordance with institutional and local regulatory requirements.
7. Needs be literate in English or native language of the country of the study enrollment to complete neuropsychological testing.
8. Subject can be reasonably expected to maintain a seizure diary alone or with the assistance of a competent individual.
9. Women of childbearing potential must be using a medically accepted method of contraception and have a negative qualitative β-human chorionic growth hormone (β-HCG) pregnancy test result from a urine or blood sample collected per SOE.

Exclusion Criteria:

* 1. Subject has any significant neurologic disease other than epilepsy. 2. Subject has had status epilepticus refractory to benzodiazepines and phenytoin in the past year 3. Subject is currently taking oral valproic acid or sodium divalproex. 4. Subject has known allergy to valproic acid, divalproex sodium, Epilim, or Depacon.

  5. Subject has unstable depression or any major psychiatric disorder including psychosis, major depression, bipolar disorder that in the opinion of the Investigator would put the subject at risk as a participant in the study.

  6. Subject has history or evidence of congestive heart failure, clinically significant peripheral edema, or anemia with a hematocrit <30%.

  7. Subject has current diagnosis of cancer requiring treatment. 8. Subject in the opinion of the Investigator, is not a suitable candidate for cranial surgery for any reason.

  9. Subject has known HIV infection or known or suspected prion disease. 10. Subject has known allergies to drugs or excipients. 11. Subject is breastfeeding, pregnant, or expressed intent on becoming pregnant during the course of the study and Investigator feels pregnancy is a likely outcome during the study 12. In the opinion of the investigator, the subject has a clinically significant or unstable medical condition (including alcohol and/or drug abuse) or a progressive CNS disease that in the opinion of the Investigator would put the subject at risk as a participant in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Safety measured as drug or device related SAEs | 2-years
  The primary objective is to assess long-term safety and tolerability of ICV delivery of Valproate as measured by drug and device related adverse events.

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (5):
  - Mater Brisbane, Brisbane, New South Wales
  - RBWH, Brisbane, New South Wales
  - SVHM, Melbourne, Victoria
  - The Alfred, Melbourne, Victoria
  - The Austin, Melbourne, Victoria
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheeba Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No